CLINICAL TRIAL: NCT03348241
Title: Randomized Controlled Trial on the Effect of Gum Arabic to Reduce Incidence of Oral Mucositis Induced by Chemotherapy for Cancer Patients
Brief Title: Using Gum Arabic for Cancer Patients to Protect From Oral Mucositis Caused by Chemotherapy: ِِِAn Experimental Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Science and Technology, Yemen (Other)
Responsible Party: Principal Investigator, Abdulrazzaq Yahya Ahmed Al Khazzan, Academic staff member, Faculty of Pharmacy, University of Science and Technology, Sana'a, Yemen., University of Science and Technology, Yemen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UST Yemen
Record Dates: First submitted 2017-11-01; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Chemotherapy-induced Oral Mucositis
Keywords: Gum Arabic; Cancer patients; Chemotherapy; Oral mucositis
MeSH Terms: conditions — Stomatitis | interventions — Gum Arabic; Drug Therapy

STUDY DESIGN:
Intervention Model Description: This is an experimental study. It was a two-arm randomized, controlled, open-label trial. The patients was categorized into two groups; study group and control group. Patients of study group was received a dose of 30 grams Gum Arabic per day as oral solution (dissolved in 250 ml purified water) for six weeks along with the chemotherapy prescribed, while patients of control group was received only chemotherapy regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gum Arabic group (Experimental): Patients of study group was received a dose of 30 grams Gum Arabic per day as oral solution (dissolved in 250 ml purified water) for six weeks along with the chemotherapy prescribed addition to verbal instructions pertaining to the optimal nutrition and daily routine for oral hygiene.
  Interventions: Drug: Gum Arabic; Drug: Chemotherapy; Behavioral: Lifestyle counseling
- Control group (Other): Patients of control group was received only chemotherapy regimen and verbal counseling pertaining to the optimal nutrition and daily routine for oral hygiene.
  Interventions: Drug: Chemotherapy; Behavioral: Lifestyle counseling

INTERVENTIONS:
Drug: Gum Arabic — Gum acacia, also known as Gum Arabic is exuded from acacia trees; mainly from Acacia Senegal (gum Hashab or Kordofan gum) which was used in this study.
  Other Names: Acacia Senegal
  Arms: Gum Arabic group
Drug: Chemotherapy — Patients of control group and study group (Gum Arabic group) received chemotherapy according to type and stage of cancer.
  Other Names: Chemotherapy agents
Behavioral: Lifestyle counseling — Lifestyle counseling pertaining to the optimal nutrition and daily routine for oral hygiene.

SUMMARY:
This study was designed to investigate the effect of Gum Arabic (GA) on cancer patients to prevent chemotherapy-induced oral mucositis. Cancer patients who will receive chemotherapy were divided into two groups; study "Gum Arabic" group (which received GA with chemotherapy) and control group (chemotherapy alone); and the participants were recruited to reach 190 patients in the study group and 184 patients in control group. This clinical trial was conducted in outpatient chemotherapy sections at Radiation and Isotopes Center of Khartoum. This study was designed to test the theory that say the chemotherapy-induced oral mucositis will significantly decrease after ingestion 30 grams as daily dose of Gum Arabic in a form of solution for six weeks during therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients whom well diagnosed with cancer in any stage were eligible for enrolment if chemotherapy is part of their treatment plan.

Exclusion Criteria: Patients were excluded if

* they had received recent previous chemotherapy or radiotherapy,
* they had oral mucositis or periodontitis,
* there is evidence of any systemic diseases.

Ages: 14 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The effect of Gum Arabic to prevent Chemotherapy-induced Oral Mucositis was the primary outcome that assessed using World Health Organization Mucositis Scoring. | Six weeks for each participant from starting therapy.
  The primary outcome measure of oral mucositis in cancer patients who received chemotherapy was depend on presence or absence oral mucositis after commencement the treatment because they were new diagnosed cases and free from oral mucositis. World Health Organization Mucositis Scale, was the scoring system used to assess oral mucositis based on a combination of subjective (soreness as described by the patient), objective (presence of erythema and ulcerations) and functional (ability to eat solids, liquids or nothing by mouth) outcomes.
  During six weeks of follow up there were specific questions that asked by researcher and had been answered by patient regarding oral mucositis. Those questions summarized as follow: 1. Does the oral mucositis was occurred during this week? 2. If Yes. Is there was soreness, erythema or ulcers in mouth of participant? 3. The day that oral mucositis was started and eliminated? 4. If the patient belong to study group; Is Gum Arabic still used regularly?

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrazzaq Y. Al khazzan, MClinPharm, Principal Investigator — University of Science and Technology

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the date that related to the time when summary data are published.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03348241/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03348241/ICF_001.pdf